CLINICAL TRIAL: NCT03295734
Title: ACES - ACE Inhibitors Combined With Exercise for Seniors With Hypertension
Acronym: ACES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Colorado, Denver (Other); AdventHealth Translational Research Institute (Other)
Responsible Party: Principal Investigator, Thomas W. Buford, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Record Dates: First submitted 2017-09-21; First posted 2017-09-28 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Aging; Sedentary Lifestyle
MeSH Terms: conditions — Hypertension; Sedentary Behavior | interventions — Exercise; Perindopril; Losartan; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Perindopril (Active Comparator): 4 mg qd titrated to 8 mg qd perindopril + aerobic exercise
  Interventions: Behavioral: Aerobic exercise; Drug: Perindopril
- Losartan (Active Comparator): 50 mg qd titrated to 100 mg qd losartan + aerobic exercise
  Interventions: Behavioral: Aerobic exercise; Drug: Losartan
- HCTZ (Active Comparator): 12.5 mg qd titrated to 25 mg qd HCTZ + aerobic exercise
  Interventions: Behavioral: Aerobic exercise; Drug: HCTZ

INTERVENTIONS:
Behavioral: Aerobic exercise — Twice weekly centered based aerobic exercise + 3/week home-based walking
Drug: Perindopril — 4 mg qd titrated to 8 mg qd perindopril
  Arms: Perindopril
Drug: Losartan — 50 mg qd titrated to 100 qd losartan
  Arms: Losartan
Drug: HCTZ — 12.5 mg qd titrated to 25 qd HCTZ
  Arms: HCTZ

SUMMARY:
The purpose of this project is to conduct a randomized, controlled trial (RCT) to determine if choice of antihypertensive medication influences changes in functional status and other cardiovascular risk factors among older persons with hypertension when combined with physical exercise.

DETAILED DESCRIPTION:
The purpose of this project is to conduct a randomized, controlled trial (RCT) to determine if choice of antihypertensive medication influences changes in functional status and other cardiovascular risk factors among older persons with hypertension. Functional status, determined by measures of physical performance, is an important predictor of cardiovascular outcomes in older adults. Seniors with compromised function experience more CV events, have a higher risk of undergoing cardiac surgery and higher risk of CVD-related death than higher-functioning peers. Seniors with hypertension experience accelerated declines in function, and presently physical exercise is the primary strategy for preventing this decline. However, functional responses to exercise are highly variable and appear to be influenced by the type of antihypertensive medication(s) utilized to control blood pressure. Preliminary evidence suggests that, compared to other first-line antihypertensive agents, angiotensin converting enzyme (ACE) inhibitors enhance exercise-derived improvements in functional status among hypertensive seniors. This RCT will test this hypothesis. Sedentary men and women > 60 years of age with functional limitations and hypertension will be recruited from two sites to participate in a longitudinal intervention study. Participants will be randomly assigned to one of three first-line antihypertensive agents: (1) the ACE inhibitor perindopril, (2) AT1 receptor antagonist losartan, or (3) the thiazide diuretic hydrochlorothiazide. Note: Participants with a documented history of hypersensitivity to ACE inhibitors will be randomized 1:1 to one of the two other study drugs. All participants will also participate in a structured aerobic exercise intervention. The primary aim is to determine if, compared to losartan and HCTZ, perindopril improves self-paced gait speed. The secondary aim is to determine the relative effect of perindopril on a) exercise capacity, b) body mass and composition, and c) circulating indices of cardiovascular risk. This study is expected to differentiate beneficial effects of three FDA-approved antihypertensive medications on an emerging cardiovascular risk factor in a clinically-relevant population. Thus the study has important implications for expeditiously influencing clinical practice guidelines in the prescription of antihypertensive drugs to millions of Americans.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and older
* Hypertension - untreated (SBP ≥ 140 mm Hg or DBP ≥ 90 mm Hg) or treated
* > 290 seconds needed to complete long-distance corridor walk test
* Sedentary lifestyle, defined as <150 min/wk of moderate physical activity
* Willingness to participate in all study procedures, including allowing study team to communicate with primary care physician regarding changes in antihypertensive treatment

Exclusion Criteria:

* BP > 140/90, despite the use of three or more anti-hypertensive drugs
* SBP > 180 mm Hg or DBP > 110 mm Hg
* Chronic kidney disease
* Serum creatinine >2.5 mg/dL in men or >2.0 mg/dL in women
* Serum potassium outside normal reference range
* Urinary protein > 1 on dipstick
* Abnormal liver enzymes (AST, ALT, or alkaline phosphatase > 2.5 times the upper limit of normal)
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Acute myocardial infarction identified by ECG
* Significant cognitive impairment, defined as a known diagnosis of dementia or a Mini-Mental State Examination exam score < 24;
* Simultaneous participation in another intervention trial
* Known hypersensitivity to ACE inhibitors (exclusion only to perindopril arm; will be randomized among other two interventions)
* Any other condition that would preclude participating based upon judgement of PI or study clinician team

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Buford, PhD, Principal Investigator — University of Alabama at Birmingham; Bret Goodpaster, PhD, Principal Investigator — Translational Research Institute, Advent Health
Locations (2):
- United States (2):
  - UAB Center for Exercise Medicine, Birmingham, Alabama
  - Translational Research Institute, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harper SA, Baptista LC, Roberts LM, Wherry SJ, Boxer RS, Hildreth KL, Seay RS, Allman PH, Carter CS, Aban I, Kohrt WM, Buford TW. Angiotensin Converting Enzyme Inhibitors Combined with Exercise for Hypertensive Seniors (The ACES Trial): Study Protocol of a Randomized Controlled Trial. Front Med (Lausanne). 2020 Jan 22;6:327. doi: 10.3389/fmed.2019.00327. eCollection 2019. PMID 32039215

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: **NOTE: Participants could be excluded for more than one reason**
  Excluded (n=274)
  • Not meeting inclusion criteria# (n=274)
  * No physical function limitation (n=107)
  * Active lifestyle (n=55)
  * Resistant hypertension (n=35)
  * Severe cardiac disease (n= 34)
  * Significant cognitive impairment (n=15)
  * No hypertension (n=13)
  * Uncontrolled hypertension (n=10)
  * Proteinuria> 1+ (n=8)
  * Other medical concern that precluded safe participation (n=65)
Period: Overall Study
Arm/Group | Perindopril | Losartan | HCTZ
Started | 74 | 74 | 75
Completed | 60 | 55 | 57
Not Completed | 14 | 19 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perindopril | Losartan | HCTZ | Total
Number analyzed (Participants) | 74 | 74 | 75 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (4.9) | 67.9 (5.8) | 67.0 (4.9) | 67.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 55 | 56 | 168
  Male | 17 | 19 | 19 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2 | 4
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 27 | 31 | 23 | 81
  White | 45 | 38 | 48 | 131
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Gait Speed From Baseline
Description: Self-paced gait speed over 4m distance; change from baseline to week 32
Time Frame: 32 weeks
Population: Intent to Treat
Measure: Mean (95% Confidence Interval); unit: m/sec
Arm/Group | Perindopril | Losartan | HCTZ
Number analyzed (Participants) | 74 | 74 | 75
m/sec | 0.10 [-0.42 to 0.61] | 0.05 [-0.43 to 0.54] | 0.10 [-.28 to 0.47]

ADVERSE EVENTS:
Time Frame: 7 months of engagement in the study
Arm/Group | Perindopril | Losartan | HCTZ
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74 | 0/75
Serious Adverse Events (participants affected / at risk) | 2/74 | 1/74 | 5/75
Other Adverse Events (participants affected / at risk) | 32/74 | 31/74 | 40/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perindopril (N=74) | Losartan (N=74) | HCTZ (N=75)
Hospitalization (General disorders) | 1 (1) | 0 (0) | 4 (4)
Other (General disorders) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perindopril (N=74) | Losartan (N=74) | HCTZ (N=75)
Musculoskeletal, muscle pulls, strains (Musculoskeletal and connective tissue disorders) | 16 | 9 | 15
Other (General disorders) | 16 | 22 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03295734/Prot_SAP_001.pdf
  • Informed Consent Form (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT03295734/ICF_002.pdf